CLINICAL TRIAL: NCT05662605
Title: A Randomized Controlled Trial of the Feasibility and Acceptability of W-PPMA for Postpartum Mothers
Brief Title: W-PPMA for Postpartum Mothers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Woebot Health (Industry)
Collaborators: Scripps Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: W-PPD-003
Record Dates: First submitted 2022-11-21; First posted 2022-12-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Period

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-PPMA (Experimental): Participants randomized to this arm will have access to the W-PPMA mobile app throughout the 16-week study. Participants are asked to use the app for at least 5 minutes a day during the treatment phase (first 8 weeks) and then as often as they like during the follow-up phase (last 8 weeks) of the study.
  Interventions: Device: W-PPMA
- Waitlist (No Intervention): Participants assigned to this group will not have access to the W-PPMA mobile app during the treatment phase (first 8 weeks) of the study. They will have access during the follow-up phase (last 8 weeks) of the study and will be instructed to use the app for at least 5 minutes a day.

INTERVENTIONS:
Device: W-PPMA — W-PPMA is a digital health tool designed specifically for the postpartum experience and is accessed through a mobile application which delivers evidence-based therapy through brief "conversations" with a fully automated relational agent called Woebot.
  Arms: W-PPMA

SUMMARY:
To evaluate the feasibility and acceptability of W-PPMA among a diverse group of postpartum mothers.

DETAILED DESCRIPTION:
This randomized waitlist-controlled trial evaluates the feasibility and acceptability of the W-PPMA digital health tool.

Participants will be recruited from the IRB-approved PowerMom research study of Scripps Research and, if interested, will complete screening for the sub-study. Eligible participants will be asked to provide informed consent and complete the baseline assessments. Those that do not meet eligibility criteria may resume their PowerMom experience.

Eligible participants will be randomized to one of two groups, W-PPMA or Waitlist, and will receive instructions on when and how they can access the digital health tool. Primary endpoints will be measured at 8-weeks (end of treatment) with additional measures being collected at 1- 4-, 8-, 12-, and 16-weeks (end of study). Screening, consenting, and outcome measures will be completed online through the MyDataHelps app.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age
* Be ≤ 3 month postpartum
* Currently enrolled in Scripps Research PowerMom study
* Own or have regular access to a smartphone (Android or iOS smartphone with a recent, supported operating system), that can receive SMS messages, and has reliable Wi-Fi access or sufficient data to engage with assigned treatment condition for the duration of the study
* Available and committed to engage with the program and complete assessments for a 16-week duration.
* Ability to read and understand English

Exclusion Criteria:

* Lifetime diagnosis of a psychotic disorder (including schizophrenia or schizoaffective disorder)
* Lifetime diagnosis of bipolar disorder
* Current suicidal ideation with a plan or intent or a suicidal attempt within the past 12 months
* History of (a) drug and/or alcohol abuse within the past 12 months
* Fetal demise within the past 18 months
* Previous use of the Woebot app

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Usage Rating Profile Intervention (URPI)-Feasibility | End of Treatment (8 weeks from baseline)
  Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Responses range from 1 = "slightly disagree" to 6 = "strongly agree". Scores are averages, with greater scores indicating greater intervention feasibility.
Usage Rating Profile Intervention (URPI)-Acceptability | End of Treatment (8 weeks from baseline)
  Measure of acceptability. A 6-item subscale that inquires about intervention acceptability. Responses range from 1 = "slightly disagree" to 6 = "strongly agree". Scores are averages, with greater scores indicating greater intervention acceptability.
Client Satisfaction Questionnaire (CSQ-8) | End of Treatment (8 weeks from baseline)
  An 8-item measure used to assess client's satisfaction with treatment on a 4-point scale (1 = "very dissatisfied" to 4 = "very satisfied"). Example questions include, "How would you rate the quality of service you received"? and "Did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with the W-PPMA mobile application.
Number of active days in the W-PPMA application | Throughout treatment (from baseline to end of treatment at 8 weeks)
  Application engagement in the total number of active days using the application will be collected during the study to provide quantitative data regarding application utilization.
Number of messages sent per week in the W-PPMA application | Throughout treatment (from baseline to end of treatment at 8 weeks)
  Application engagement in the number of messages sent each week within the application will be collected during the study to provide quantitative data regarding application utilization.
Number of modules completed in the W-PPMA application | Throughout treatment (from baseline to end of treatment at 8 weeks)
  Application engagement in the number of modules completed within the application will be collected during the study to provide quantitative data regarding application content engagement.
Content satisfaction ratings in the W-PPMA application | Throughout treatment (from baseline to end of treatment at 8 weeks)
  Application content satisfaction ratings will be collected during the study to provide quantitative data regarding application content engagement.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | Change from Baseline to End of Treatment at 8 weeks)
  An 8-item abbreviated version of the PHQ-9 used to assess mood and anxiety symptoms respectively. The PHQ-8 excludes an item assessing suicidality. Total score between 0-27, where higher scores indicate greater levels of depression.
Edinburgh Prenatal Depression Scale (EPDS) | Change from Baseline to End of Treatment at 8 weeks
  A 10-item self-report questionnaire used as a screening tool to identify patients who are at risk for perinatal depression. The scale assesses depression criteria including anhedonia, worry, and sleep disturbance, in the past seven days. Each item has four ordinal response options, yielding a total score of 0 to 30 such that higher scores indicate more severe symptoms.
Generalized Anxiety Disorder Questionnaire (GAD-7) | Change from Baseline to End of Treatment at 8 weeks
  A 7-item brief self-report measure used to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. Total score between 0-21, where higher scores indicate greater levels of anxiety.
Perceived Stress Scale (PSS-10) | Change from Baseline to End of Treatment at 8 weeks
  A 10-item self-reported questionnaire designed to measure the degree to which situations in one's life are appraised as stressful. Items comprising the PSS-10 assess the frequency of experiencing certain thoughts and feelings (e.g., feelings of upset, nervousness, a lack of control) over the past month. Each item is scored on a 5-point Likert scale from 0 (never) to 4 (very often); four positively stated items are reverse scored before summing all items to obtain the total score. Higher PSS scores indicate greater perceived stress.

OTHER OUTCOMES:
Mother Infant Bonding Scale (MIBS) | Change from Baseline to End of Treatment at 8 weeks
  The MIBS consists of 8 one-word items describing an emotional response, such as ''loving'', "resentful", and ''disappointed" and is designed to assess the feelings of a mother toward her new baby. Mothers rate the degree to which they feel each of the 8 emotional responses toward their infant using a 4-point Likert scale from very much (0) to not at all (3). Five items describe negative emotional responses and are reverse scored. Total scores can range from 0 to 24, with lower scores indicating better bonding.
Working Alliance Inventory (WAI-SR) | Day 3 and End of Treatment at 8 weeks
  A validated 12-item instrument that measures therapeutic alliance. The instrument consists of a composite score and three subscales assessing key aspects of the therapeutic alliance: 1) agreement between the client and therapist on the tasks of therapy (e.g., "As a result of these sessions I am clearer as to how I might be able to change"); 2) agreement between the client and therapist on the goals of therapy (e.g., "Woebot and I collaborate on setting goals for my therapy"), and 3) the development and strength of an affective bond between the client and therapist (e.g., "Woebot and I respect each other"). The WAI-SR will be tailored to the current intervention, replacing the term "therapist" with "Woebot".
Feasibility, acceptability, perceptions of stigma as a barrier to mental health care, and mood outcomes across key sociodemographic variables of race and ethnicity, age, and level of education | Baseline, Day 3 and End of Treatment at 8 weeks
  Named outcome measures will be descriptively characterized and results will be stratified according to race and ethnicity, age group, and level of education.

CONTACTS AND LOCATIONS:
Overall Officials: Lase Ajayi, MD, Principal Investigator — Scripps Research Translational Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No